CLINICAL TRIAL: NCT03365765
Title: Exploratory Study on the Efficacy and the Safety of mFOLFOX6 Chemotherapy With Apatinib as Postoperative Treatment in Stage IIIB or IIIC Colorectal Cancer
Brief Title: mFOLFOX6 Chemotherapy With Apatinib as Postoperative Treatment in Stage IIIB or IIIC Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianbin Xiang, professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2017-299
Record Dates: First submitted 2017-11-23; First posted 2017-12-07 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Apatinib
MeSH Terms: interventions — apatinib; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This study has one Intervention Type of Drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOX6 & apatinib (Experimental): oxaliplatin 85mg/m2 intravenous infusion for 2 hours, intravenous infusion of leucovorin 400mg/m2 for 2 hours, intravenous infusion of 5- fluorouracil 400mg/m2, first days; 5- fluorouracil 2400mg/m2 continuous intravenous infusion for 46-48 hours, repeated 1 time every two weeks, a total of 12 cycles, 24 weeks. Patients also take apatinib, 1 time daily, 500mg each time, lasting 1 year, from the first chemotherapy of mFOLFOX6.
  Interventions: Drug: Apatinib; Drug: Oxaliplatin; Drug: 5-fluorouracil
- mFOLFOX6 (Active Comparator): oxaliplatin 85mg/m2 intravenous infusion for 2 hours, intravenous infusion of leucovorin 400mg/m2 for 2 hours, intravenous infusion of 5- fluorouracil 400mg/m2, first days; 5- fluorouracil 2400mg/m2 continuous intravenous infusion for 46-48 hours, repeated 1 time every two weeks, a total of 12 cycles, 24 weeks.
  Interventions: Drug: Oxaliplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Apatinib — Apatinib tablet
  Other Names: YN968D1
  Arms: mFOLFOX6 & apatinib
Drug: Oxaliplatin — Oxaliplatin Intravenous
  Other Names: Eloxatin
Drug: 5-fluorouracil — 5-fluorouracil Intravenous
  Other Names: Adrucil, Carac, Efudex, Efudix

SUMMARY:
This study will focus on postoperative patients of stage IIIB or stage IIIC colorectal cancer. These patients will start to accept chemotherapy in 3-4 weeks after operation, these patients were randomly divided into two groups, one group will accept adjuvant chemotherapy of mFOLFOX6; another group will use mFOLFOX6 combined with apatinib. The efficacy and safety of adjuvant chemotherapy will be compared between the two groups. Disease-free survival, overall survival, incidence of adverse reaction of chemotherapy and postoperative quality of life will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent form;
2. confirmed as colorectal cancer by pathology, and the stage is IIIB /IIIC according to the NCCN guidelines;
3. patients with primary colorectal cancer;
4. radical resection of colon cancer (CME) or radical resection of rectal cancer (TME) has done;
5. 3~4 weeks after radical resection ;
6. patients did not receive any radiotherapy and chemotherapy before operation

Exclusion Criteria:

1. emergency operation for colorectal cancer patients;
2. the situation after operation can not tolerance for systemic adjuvant chemotherapy (hemoglobin <95g/L, white blood cell <3 * 109/L, granulocyte <1.5 * 109/L and platelet <75 * 109/L, bilirubin>2.5N, alanine aminotransferase >2.5N, alkaline phosphatase >2.5N, urea nitrogen >2.5N, creatinine >2.5N, proteinuria, hematuria, temperature of >38 degree);
3. serious diseases such as cardiac insufficiency, respiratory insufficiency, liver and kidney dysfunction, serious blood diseases;
4. patients participated in other clinical trials at the same time;
5. pregnant or perinatal women;
6. combined with other malignant tumors;
7. a history of neuropsychiatric disorders;
8. patients have used anti angiogenesis targeted drugs (such as bevacizumab, cetuximab);
9. patients had a history of severe trauma within 4 weeks before admission;
10. allergic to chemotherapy drugs or apatinib;
11. active bleeding, ulcers, intestinal perforation, intestinal obstruction, hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 5 years
  observe the recurrence of colorectal cancer after operation

SECONDARY OUTCOMES:
overall survival | 5 years
  observe the postoperative survival rate in patients with stage IIIB and IIIC colorectal cancer
incidence of adverse reactions after chemotherapy | one year
  observe the adverse reaction of apatinib or combined chemotherapy using apatinib

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
our study protocol,statistical analysis plan,informed consent form and clinical study report are Chinese.

REFERENCES:
- [Result] Scott AJ, Messersmith WA, Jimeno A. Apatinib: a promising oral antiangiogenic agent in the treatment of multiple solid tumors. Drugs Today (Barc). 2015 Apr;51(4):223-9. doi: 10.1358/dot.2015.51.4.2320599. PMID 26020064
- [Result] Mi YJ, Liang YJ, Huang HB, Zhao HY, Wu CP, Wang F, Tao LY, Zhang CZ, Dai CL, Tiwari AK, Ma XX, To KK, Ambudkar SV, Chen ZS, Fu LW. Apatinib (YN968D1) reverses multidrug resistance by inhibiting the efflux function of multiple ATP-binding cassette transporters. Cancer Res. 2010 Oct 15;70(20):7981-91. doi: 10.1158/0008-5472.CAN-10-0111. Epub 2010 Sep 28. PMID 20876799
- [Result] Tong XZ, Wang F, Liang S, Zhang X, He JH, Chen XG, Liang YJ, Mi YJ, To KK, Fu LW. Apatinib (YN968D1) enhances the efficacy of conventional chemotherapeutical drugs in side population cells and ABCB1-overexpressing leukemia cells. Biochem Pharmacol. 2012 Mar 1;83(5):586-97. doi: 10.1016/j.bcp.2011.12.007. Epub 2011 Dec 16. PMID 22212563
- [Result] Tian S, Quan H, Xie C, Guo H, Lu F, Xu Y, Li J, Lou L. YN968D1 is a novel and selective inhibitor of vascular endothelial growth factor receptor-2 tyrosine kinase with potent activity in vitro and in vivo. Cancer Sci. 2011 Jul;102(7):1374-80. doi: 10.1111/j.1349-7006.2011.01939.x. Epub 2011 May 9. PMID 21443688
- [Result] Willett CG, Boucher Y, di Tomaso E, Duda DG, Munn LL, Tong RT, Chung DC, Sahani DV, Kalva SP, Kozin SV, Mino M, Cohen KS, Scadden DT, Hartford AC, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Chen HX, Shellito PC, Lauwers GY, Jain RK. Direct evidence that the VEGF-specific antibody bevacizumab has antivascular effects in human rectal cancer. Nat Med. 2004 Feb;10(2):145-7. doi: 10.1038/nm988. Epub 2004 Jan 25. PMID 14745444